CLINICAL TRIAL: NCT03865173
Title: Post-stroke Pathway: Analysis and Link With One Year Sequelae in a French Cohort of Stroke Patients
Acronym: PAPASéPA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/30
Record Dates: First submitted 2019-02-22; First posted 2019-03-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Stroke Sequelae
Keywords: Stroke; Pathways; Sequelae; Health services research
MeSH Terms: conditions — Stroke | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Telephone Interview — Telephone Interview

SUMMARY:
The link between post-stroke pathways and patient sequelae have not yet been clearly defined. The main purpose is to identify the post-stroke life pathways components associated with sequalae at 3 months and 1 year after the acute stroke episode.

DETAILED DESCRIPTION:
Stroke is a serious health event, involving the entire health care system and generating considerable socioeconomic weight for society. Knowledge of the components, the diversity and the scalability of post-stroke life pathways is currently not sufficient. Moreover the link between post-stroke pathways and patient sequelae have not yet been clearly defined.

The main purpose is to identify the post-stroke life pathways components associated with sequalae at 3 months and 1 year after the acute stroke episode. The secondary objectives are: 1) To define a typology of the life pathways of stroke patients, , 2) To analyze the social and geographical inequalities in the management of stroke, 4) To estimate the cost of the pathway elements of stroke management; 5) Measure the sequelae of stroke patients at three months and one year after the acute episode.

The design is a prospective multicenter cohort study with a follow up to 1 year after the acute episode, managed in several hospitals in the Aquitaine region (France).

ELIGIBILITY:
Inclusion Criteria:

* Patient being over 18 years of age living in metropolitan France;
* Patient with recent stroke (not before 2019) whose diagnosis confirmed by a neuro-vascular physician;
* Patient managed for stroke in one of the 13 participating hospitals of the Aquitaine region;
* Patient giving consent to participate to PAPASéPA;
* Patient to be alive at the end of the acute management hospital stay

Exclusion Criteria:

* Patient refuse to participate to PAPASéPA
* Patient died during the initial stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a confirmed ischemic or hemorrhagic stroke included in the Aquitaine Observatory of Stroke (ObA2) cohort and managed in the 13 participants centers and voluntary to participate
Sampling Method: Probability Sample
Enrollment: 1138 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-11-18 (Estimated); Study Completion 2022-11-18 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) Score | 3 months
  Activity limitations post-stroke measure. Minimum score : 0 "No symptoms at all " Maximum score : 6 "Dead"
Modified Rankin Scale (mRS) Score | 1 year
  Activity limitations post-stroke measure Minimum score : 0 "no symptom" Maximum score : 6 "death"

SECONDARY OUTCOMES:
Telephone Interview for Cognitive Status Modified (TICS) Score | 3 months
  Cognitive disorders post-stroke measure Score from 0 to 43
Telephone Interview for Cognitive Status Modified (TICS) Score | 1 year
  Cognitive disorders post-stroke measure Score from 0 to 43
Hospital anxiety and depression scale (HADS) Score | 3 months
  Depression and anxiety disorders post-stroke measure Scores ranged from 0 (minimum) to 21 (maximum) for anxiety and 0 (minimum) to 21 (maximum) for depression.
  Total score from 0 to 42
Hospital anxiety and depression scale (HADS) Score | 1 year
  Depression and anxiety disorders post-stroke measure Scores ranged from 0 (minimum) to 21 (maximum) for anxiety and 0 (minimum) to 21 (maximum) for depression.
  Total score from 0 to 42
Fatigue Severity Scale (FSS) Score | 3 months
  The Fatigue Severity Scale (FSS) is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. Essentially, the FSS consists of answering a short questionaire that requires the subject to rate his or her own level of fatigue. The subject is asked to read each statem ent and circle a number from 1 to 7, depending on how appropriate they felt the statement applied to them over the preceding week. A low value indicates that the statement is not very appropriate whereas a high value indicates agreement. The scoring is done by calculating the average response to the questions (adding up all the answers and dividing by nine).
  People with depression alone score about 4.5. People with fatigue average about 6.5.
Fatigue Severity Scale (FSS) Score | 1 year
  The Fatigue Severity Scale (FSS) is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. Essentially, the FSS consists of answering a short questionaire that requires the subject to rate his or her own level of fatigue. The subject is asked to read each statem ent and circle a number from 1 to 7, depending on how appropriate they felt the statement applied to them over the preceding week. A low value indicates that the statement is not very appropriate whereas a high value indicates agreement. The scoring is done by calculating the average response to the questions (adding up all the answers and dividing by nine).
  People with depression alone score about 4.5. People with fatigue average about 6.5.
Barthel Index (BI) Score | 3 months
  Functional outcome post-stroke measure The original 10-item form of the BI consists of 10 common ADL activities including: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Items are rated in terms of whether individuals can perform activities independently, with some assistance, or are dependent (scored as 10, 5 or 0). Items are weighted according to the level of nursing care required.
  Total score from 0 to 100
Barthel Index (BI) Score | 1 year
  Functional outcome post-stroke measure The original 10-item form of the BI consists of 10 common ADL activities including: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Items are rated in terms of whether individuals can perform activities independently, with some assistance, or are dependent (scored as 10, 5 or 0). Items are weighted according to the level of nursing care required.
  Total score from 0 to 100
Community Integration Questionnaire (CIQ-R) Score | 3 months
  Participation restrictions post-stroke measure Score from 0 to 35
Community Integration Questionnaire (CIQ-R) Score | 1 year
  Participation restrictions post-stroke measure Score from 0 to 35

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CH Agen, Agen
  - CH Blaye, Blaye
  - CHU Bordeaux, Bordeaux
  - CH Arcachon, La Teste-de-Buch
  - CH Sud Gironde - Langon, Langon
  - Clinique Mutualiste Lesparre Médoc, Lesparre-Médoc
  - CH Libourne, Libourne
  - CHIC Marmande-Tonneins, Marmande
  - CH Mont de Marsan - site Layné, Mont-de-Marsan
  - CH Oloron, Oloron-Sainte-Marie
  - CH Orthez, Orthez
  - CH Pau, Pau
  - Pôle de Santé du Villeneuvois, Villeneuve-sur-Lot

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broussy S, Rouanet F, Lesaine E, Domecq S, Kret M, Maugeais M, Aly F, Dehail P, Benard A, Wittwer J, Salamon R, Sibon I, Saillour-Glenisson F. Post-stroke pathway analysis and link with one year sequelae in a French cohort of stroke patients: the PAPASePA protocol study. BMC Health Serv Res. 2019 Oct 29;19(1):770. doi: 10.1186/s12913-019-4522-2. PMID 31665006